CLINICAL TRIAL: NCT00480571
Title: An Open-label, Multi-center, 6-week, Sequential Cohort Study Designed to Determine the Safety and Tolerability of Two Dose Ranges of BL-1020 in Hospitalized Subjects With Chronic Schizophrenia or Schizo-affective Disorder
Brief Title: Safety and Tolerability of BL-1020 in Hospitalized Subjects With Chronic Schizophrenia or Schizo-Affective Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: BioLineRx, Drug Development Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-1020 II
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2007-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: chronic schizophrenia or schizo-affective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — perphenazine GABA ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): BL 1020 low dose
  Interventions: Drug: BL-1020
- 2 (Experimental): BL 1020 High Dose
  Interventions: Drug: BL 1020 High Dose

INTERVENTIONS:
Drug: BL-1020 — BL-1020 Low Dose
  Arms: 1
Drug: BL 1020 High Dose — BL 1020 High Dose
  Arms: 2

SUMMARY:
An open-label, multi-center, 6-week, sequential cohort study designed to determine the safety and tolerability of two dose ranges of BL-1020 in hospitalized subjects with chronic schizophrenia or schizo-affective disorder

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 to 65 years of age, inclusive
* meet criteria for chronic (diagnosis established > 1 year ago) schizophrenia with adequate psychotic symptoms as demonstrated by a PANSS total score > 60
* current diagnosis of schizophrenia (disorganized type, 295.10; catatonic type, 295.20; paranoid type, 295.30; undifferentiated type, 295.90) or schizoaffective disorder (295.7) in accordance with DSM-IV
* Agree to be fully hospitalized until at least Day 14 of the study
* Females must be of non-childbearing potential: surgically sterilized (i.e. tubal ligation), have had a hysterectomy prior to the screening phase, or be post-menopausal. Females who have been post-menopausal for more than 12 months but less than 24 months must have a FSH > 40 mU/mL.

Exclusion Criteria:

* Pregnant or lactating women
* administration of clozapine within 60 days prior to Baseline
* DSM-IV diagnosis of schizophreniform disorder (295.40) or schizophrenia residual sub-type (295.60), or other primary psychiatric diagnoses, such as bipolar disorder or major depressive disorder
* Severity of psychosis rated severe or higher (CGI-S 6 or 7)
* Known suicidal risk (modified ISST score>7)
* Requiring disallowed concomitant psychotropic medication following enrolment into the study
* Current evidence of clinically significant or unstable illness
* Clinically significant abnormal laboratory data (e.g. creatinine, AST or ALT greater than 3 x the upper limit of normal, TSH>10 IU) at screening, or any abnormal laboratory values that could interfere with the assessment of safety (e.g. blood cell count, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of two dose ranges (20-40 mg/day, 30-50 mg/day) of BL-1020 tri-mesylate (free base) in subjects with chronic schizophrenia or schizo-affective disorder | 6 weeks

SECONDARY OUTCOMES:
To determine the MTD, the optimal dose escalation schedule, and the maximum tolerated maintenance dose | 6 weeks
To compare the efficacy of the two dose ranges of BL-1020 | 6 weeks
To determine the pharmacokinetics of BL-1020 and its metabolites | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davidson, MD, Principal Investigator — Dept. of Psychiatry, Sheba Medical Center
Locations (2):
- Dept. of Psychiatry, Sheba Medical Center, Tel Litwinsky, Israel
- Spitalul Clinic de Urgenţǎ Militar Central "Dr Carol Davila",, Bucharest, Str Mircea Vulcǎnescu 18, Romania